CLINICAL TRIAL: NCT05009602
Title: Diagnostic Tools to Establish the Presence and Severity of Peripheral Arterial Disease in People With Diabetes
Acronym: DM PAD
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Leicester (Other); University of Edinburgh (Other); Universidad de Granada (Other)
Responsible Party: Sponsor
Other Study IDs: 21CX7046
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot; Peripheral Arterial Disease; Diabetic Foot Ulcer; Peripheral Vascular Diseases; Peripheral Artery Disease; Critical Limb Ischemia; Critical Lower Limb Ischemia
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Ankle Brachial Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participating Centre: To complete all index tests and reference scan
  Interventions: Diagnostic Test: Toe Brachial Pressure Index (TBPI); Diagnostic Test: Ankle Brachial Pressure Index (ABPI); Diagnostic Test: Exercise Ankle Brachial Pressure Index (ABPI); Diagnostic Test: Audible handheld Doppler; Diagnostic Test: Visual handheld Doppler; Diagnostic Test: Podiatry Ankle Duplex scan (PAD-scan)

INTERVENTIONS:
Diagnostic Test: Toe Brachial Pressure Index (TBPI) — TBPI will be measured using the photoplethysmography (PPG) method, employing an infrared sensor placed on the hallux and index finger.
Diagnostic Test: Ankle Brachial Pressure Index (ABPI) — A sphygmomanometer-cuff placed at the ankle and a handheld continuous wave Doppler device will be used to measure the systolic pressure of the dorsalis pedis and posterior tibial artery.
Diagnostic Test: Exercise Ankle Brachial Pressure Index (ABPI) — A sphygmomanometer-cuff placed at the ankle and a handheld continuous wave Doppler device will be used to measure the systolic pressure of the dorsalis pedis and posterior tibial artery, following the participant completing 50 consecutive repetitions of active dorsiflexion whilst standing.
Diagnostic Test: Audible handheld Doppler — Audible CW Doppler interrogation of the dorsalis pedis and posterior tibial artery.
Diagnostic Test: Visual handheld Doppler — Visual CW interrogation of the dorsalis pedis and posterior tibial artery was performed using the handheld Huntleigh Digital Dopplex device.
Diagnostic Test: Podiatry Ankle Duplex scan (PAD-scan) — Podiatry ankle duplex scan (PAD-scan) involves using an ultrasound machine to visualise the anterior and posterior tibial arteries at the ankle.
  To be used in 3 participating centers only.

SUMMARY:
In the UK there are over 7,000 leg amputations each year because of diabetes. The most important cause of this is poor circulation. The detection of poor circulation in patients with diabetes is difficult. A number of tests exist to detect poor circulation (known as peripheral arterial disease (PAD)). However, there is confusion as to which is the gold standard.

The DM PAD study aims to determine the diagnostic performance of index tests (audible handheld Doppler, visual handheld Doppler, ankle brachial pressure index (ABPI), exercise ABPI and toe brachial pressure index (TBPI)) for the diagnosis of PAD in patients with diabetes as determined by a reference test (CTA or MRA).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Known history of diabetes

Exclusion Criteria:

* PAD status known on imaging
* Known history of PAD intervention
* CTA and MRA contraindications- renal impairment, pregnancy, contrast medium hypersensitivity/allergy, non-compatible implants (MRA only).
* Unable to provide appropriate informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usman Jaffer, Principal Investigator — Chief Investigator
Locations (17):
- United Kingdom (17):
  - Mid and South Essex NHS Foundation Trust, Basildon
  - Cardiff and Vale UHB, Cardiff
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - NHS Greater Glasgow and Clyde, Glasgow
  - Hull University Teaching Hospitals NHS Trust, Hull
  - University Hospitals of Leicester NHS Trust, Leicester
  - Central London Community Healthcare NHS Trust sites, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Hammersmith and Fulham Partnership, London
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Nottingham University Hospitals (NUH) NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - University Hospitals Southampton NHS Foundation Trust, Southampton
  - Worcestershire Acute Hospitals NHS Trust, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Normahani P, Burgess L, Norrie J, Epstein DM, Kandiyil N, Saratzis A, Smith S, Khunti K, Edmonds M, Ahluwalia R, Coward T, Hartshorne T, Ashwell S, Shalhoub J, Pigott E, Davies AH, Jaffer U; DM PAD study investigators. Study protocol for a multicentre comparative diagnostic accuracy study of tools to establish the presence and severity of peripheral arterial disease in people with diabetes mellitus: the DM PAD study. BMJ Open. 2022 Nov 3;12(11):e066950. doi: 10.1136/bmjopen-2022-066950. PMID 36328388

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients are assessed for eligibility and some are excluded as per eligibility criteria
Groups:
- All Participants: Diagnostic Test: Toe Brachial Pressure Index (TBPI) TBPI will be measured using the photoplethysmography (PPG) method, employing an infrared sensor placed on the hallux and index finger.
  Diagnostic Test: Ankle Brachial Pressure Index (ABPI) A sphygmomanometer-cuff placed at the ankle and a handheld continuous wave Doppler device will be used to measure the systolic pressure of the dorsalis pedis and posterior tibial artery.
  Diagnostic Test: Exercise Ankle Brachial Pressure Index (ABPI) A sphygmomanometer-cuff placed at the ankle and a handheld continuous wave Doppler device will be used to measure the systolic pressure of the dorsalis pedis and posterior tibial artery, following the participant completing 50 consecutive repetitions of active dorsiflexion whilst standing.
  Diagnostic Test: Audible handheld Doppler Audible CW Doppler interrogation of the dorsalis pedis and posterior tibial artery.
  Diagnostic Test: Visual handheld Doppler Visual CW interrogation of the dorsalis pedis and posterior tibial artery was performed using the handheld Huntleigh Digital Dopplex device.
  Diagnostic Test: Podiatry Ankle Duplex scan (PAD-scan) Podiatry ankle duplex scan (PAD-scan) involves using an ultrasound machine to visualise the anterior and posterior tibial arteries at the ankle.
  To be used in 3 participating centers only.
Period: Overall Study
Arm/Group | All Participants
Started | 604
Completed | 536
Not Completed | 68

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for 603 participants that underwent baseline index tests
Arm/Group | All Participants
Number analyzed (Participants) | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.48 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215
  Male | 388
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 429
  Asian | 83
  Black | 47
  Mixed race / multiple ethnic background | 12
  Other ethnic group | 31
  Missing | 1
Diabetes mellitus type [Count of Participants; unit: Participants]
  Type 1 | 115
  Type 2 | 480
  Missing | 8
Previous history of diabetic foot ulcer [Count of Participants; unit: Participants]
  Yes | 68
  No | 595
Leg pain at rest [Count of Participants; unit: Participants]
  Yes | 165
  No | 438
Leg pain whilst exercising [Count of Participants; unit: Participants]
  Yes | 157
  No | 446
Gangrene [Count of Participants; unit: Participants]
  Yes | 8
  No | 595
Foot examination - ulceration [Count of Participants; unit: Participants]
  Yes | 82
  No | 521
Foot examination - Infection [Count of Participants; unit: Participants]
  Yes | 27
  No | 576
Foot examination - Neuropathy present in index limb [Count of Participants; unit: Participants]
  Yes | 148
  No | 455
Overall WIfI Score [Count of Participants; unit: Participants] — Foot examination (neuropathy, pedal pulse examination, presence of diabetic foot ulcer (DFU), DFU severity using the WIfI (Wound, Ischemia, foot Infection) classification system.
  Categories are very low, low, moderate and high - referring to the risk of amputation at 1 year.
  Participants
    Very Low | 564
    Low | 13
    Moderate | 16
    High | 3
    Missing | 7

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy of the PAD-scan and other bedside tests will be compared to the results of a Magnetic resonance angiograph (MRA) or Computed tomography angiography (CTA) (reference test).
Time Frame: 6 weeks; all index tests will be performed on the same day of presentation; reference scan performed within six weeks of the index tests.
Population: Number of participants who underwent the index test
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Audible Doppler: Audible CW Doppler interrogation of the dorsalis pedis and posterior tibial artery.
- Visual Doppler: Visual CW interrogation of the dorsalis pedis and posterior tibial artery was performed using the handheld Huntleigh Digital Dopplex device.
- Podiatry Ankle Duplex Scan (PAD-scan): Podiatry ankle duplex scan (PAD-scan) involves using an ultrasound machine to visualise the anterior and posterior tibial arteries at the ankle.
  Used in 3 participating centers only.
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | Podiatry Ankle Duplex Scan (PAD-scan)
Number analyzed (Participants) | 536 | 536 | 521 | 532 | 480 | 101
percentage
  Sensitivity | 36 [27 to 45] | 42 [33 to 51] | 55 [46 to 64] | 41 [32 to 50] | 41 [31 to 51] | 89 [74 to 100]
  Specificity | 93 [90 to 97] | 86 [81 to 91] | 78 [72 to 83] | 84 [79 to 89] | 83 [78 to 88] | 69 [54 to 84]
  Positive Predictive Value (PPV) | 75 [64 to 87] | 63 [52 to 74] | 58 [48 to 67] | 59 [48 to 70] | 55 [44 to 67] | 57 [38 to 76]
  Negative Predictive Value (NPV) | 72 [66 to 77] | 72 [66 to 78] | 76 [70 to 81] | 71 [66 to 77] | 74 [68 to 80] | 93 [84 to 100]

2. Primary Outcome: Diagnostic Accuracy - Ratios
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Number of participants who underwent the index test
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | Podiatry Ankle Duplex Scan (PAD-scan)
Number analyzed (Participants) | 536 | 536 | 521 | 532 | 480 | 101
ratio
  Negative Likelihood Ratio (NLR) | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.8] | 0.6 [0.5 to 0.7] | 0.7 [0.6 to 0.8] | 0.7 [0.6 to 0.8] | 0.2 [0.0 to 0.6]
  Positive Likelihood Ratio (PLR) | 5.3 [3.0 to 9.4] | 3.0 [2.0 to 4.5] | 2.5 [1.8 to 3.4] | 2.6 [1.7 to 3.8] | 2.4 [1.6 to 3.6] | 2.9 [1.7 to 4.9]
  Odds Ratio (OR) | 7.7 [3.9 to 15.1] | 4.4 [2.5 to 7.6] | 4.2 [2.5 to 7.0] | 3.7 [2.1 to 6.3] | 3.4 [2.0 to 6.1] | 18.8 [3.4 to 106]

3. Secondary Outcome: Health Economic Outcome - Cost Effectiveness
Description: Incremental cost-effectiveness ratio at 5 years.
Time Frame: 5 years
Population: The costs over 5 years for a hypothetical cohort of 1000 diabetic patients that is similar to the DM PAD cohort.
  Weighted average costs.
Measure: Mean (95% Confidence Interval); unit: GBP
Groups:
- No Test: "No test" supposes a scenario where diabetic patients are offered neither bedside tests nor DUS, and receive usual care for non-PAD diabetic patients.
- DUS for All: DUS for all considers a scenario where all diabetic patients are offered anatomical imaging at baseline, without a previous bedside test.
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | No Test | DUS for All
Number analyzed (Participants) | 1000 | 1000 | 1000 | 1000 | 1000 | 1000 | 1000
GBP
  Cost (£) | 11165437 [10346360 to 12197728] | 11204467 [10244720 to 12440400] | 11241003 [10057894 to 12,905,315] | 11218496 [10272695 to 12476374] | 11229209 [10328808 to 12502669] | 11156745 [11156745 to 11156745] | 11413487 [9190648 to 14285664]
  Net benefit (£) | 37186446 [35752535 to 38475241] | 37310327 [35587599 to 38724440] | 37607662 [35404894 to 39371581] | 37273035 [35626018 to 38725778] | 37267357 [35554592 to 38677467] | 36240553 [36240553 to 36240553] | 38641671 [34660841 to 41716288]

4. Secondary Outcome: Health Economic Outcome - Cost Effectiveness (QALY)
Description: Incremental cost-effectiveness ratio at 5 years.
Time Frame: 5 years
Population: Hypothetical cohort of 1000 diabetic patients that is similar to the DM PAD cohort
Measure: Mean (95% Confidence Interval); unit: Quality Adjusted Life Years
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | No Test | DUS for All
Number analyzed (Participants) | 1000 | 1000 | 1000 | 1000 | 1000 | 1000 | 1000
Quality Adjusted Life Years | 2418 [2392 to 2448] | 2426 [2397 to 2454] | 2442 [2407 to 2477] | 2425 [2397 to 2453] | 2425 [2397 to 2455] | 2370 [2370 to 2370] | 2503 [2444 to 2548]

5. Secondary Outcome: Patient Acceptability
Description: Patients will be asked to rate their experience of each index test on a Likert scale.
Time Frame: 1 hour: all index tests will be performed on the same day of presentation.
Population: Participant that underwent the index test
Measure: Number; unit: participants
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | Podiatry Ankle Duplex Scan (PAD-scan)
Number analyzed (Participants) | 603 | 603 | 603 | 603 | 603 | 101
participants
  Very unsatisfied | 7 | 7 | 7 | 11 | 8 | 2
  Unsatisfied | 1 | 1 | 0 | 6 | 6 | 0
  Neutral | 6 | 5 | 6 | 13 | 12 | 2
  Satisfied | 84 | 81 | 81 | 89 | 77 | 21
  Very satisfied | 501 | 503 | 494 | 475 | 435 | 77
  Missing | 4 | 6 | 15 | 9 | 65 | 0

6. Secondary Outcome: Technical Success
Description: Inability to perform, refusal and discontinuation of tests will be documented
Time Frame: as for outcome 1
Population: Recruited participants
Measure: Count of Participants; unit: Participants
Arm/Group | Audible Doppler | Visual Doppler | Toe Brachial Pressure Index (TBPI) | Ankle Brachial Pressure Index (ABPI) | Exercise Ankle Brachial Pressure Index (ABPI) | Podiatry Ankle Duplex Scan (PAD-scan)
Number analyzed (Participants) | 603 | 603 | 603 | 603 | 603 | 103
Participants
  Assessment performed - yes | 603 | 603 | 590 | 599 | 540 | 102
  Assessment performed - no | 0 | 0 | 13 | 4 | 63 | 1
  Assessment discontinued - yes | 0 | 0 | 4 | 3 | 7 | 0
  Assessment discontinued - no | 603 | 603 | 586 | 596 | 533 | 102

ADVERSE EVENTS:
Time Frame: Reported during the study duration; approximately 6 weeks (from baseline until scan performed).
Description: An AE is any untoward medical occurrence in a patient or clinical trial participant. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, whether or not considered related to the trial protocol.
  For the purposes of the study, only AEs related to study procedures were recorded.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/604
Serious Adverse Events (participants affected / at risk) | 0/604
Other Adverse Events (participants affected / at risk) | 4/604
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=604)
Bilateral Leg pain (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) — Patient vomited after completing exercise ABPI
Cramp and leg pain (Vascular disorders) | 1 (1) — Cramp and leg pain after first visit
Leg pain (Vascular disorders) | 1 (1) — Participant complained of left lower leg pain and leg 'occasionally giving way' for five days following index tests. Reports nothing since

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT05009602/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT05009602/SAP_001.pdf